CLINICAL TRIAL: NCT02994992
Title: Sun Protection Factor (SPF) Assay: UVA Protection Factor Assay Minimal Persistent Pigment-Darkening Dose
Brief Title: Sun Protection Factor Assay (316/2016)
Acronym: SPF Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19316
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF evaluation (Experimental): Each test site area is divided into test sub site areas that are approximately at least 0.5 cm*2. The application of test material is 2 mg/cm*2. Thus, each 50 cm*2 test site area of a subject requires 100 mg of a test material to obtain a standard 2 mg/cm*2 test application.
  Interventions: Drug: BAY 987516; Drug: SPF Control

INTERVENTIONS:
Drug: BAY 987516 — Each 50 cm*2 test site area of a subject requires 100 mg of a test material to obtain a standard 2 mg/cm*2 test application. (Formulation Code: Z46-100)
Drug: SPF Control — Each 50 cm*2 test site area of a subject requires 100 mg of a test material to obtain a standard 2 mg/cm*2 test application.

SUMMARY:
To evaluate the Sun Protection Factor efficacy on human skin.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type l, ll and/or lll for UVB testing. Fitzpatrick Skin Type ll, lll and/or lV for UVA testing.
* Male and female.
* Aged between 18-70 years old.
* Good health as determined from the HRL SHF (Subject History Form).
* Signed and dated Informed Consent Form
* Signed and dated HIPAA (Health Insurance Portability and Accountability Act) form.
* An unambiguous MED (Minimal Erythema Dose) or MPPD (Minimal Persistent Pigment Darkening Dose).

Exclusion Criteria:

* Subjects on test at any other research laboratory or clinic.
* Known allergy or sensitivity to sunscreens, cosmetics and toiletries, topical drugs and/or ultraviolet light.
* Pre-existing dermatologic conditions which have been diagnosed by a medical professional (e.g. psoriasis, eczema, etc.) which would interfere with this study.
* Pre-existing other medical conditions (e.g. adult asthma, diabetes).
* Treatment with antihistamines or corticosteroids within one week prior to initiation of the test.
* Treatment with antibiotics within two weeks prior to initiation of the test.
* Chronic medication which could affect the results of the study.
* Known pregnant or nursing women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
Minimal Erythema Dose (MED) | Up to 15 minutes
Minimal Persistent Pigment Darkening Dose (MPPD) | Up to 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Union, New Jersey, United States